CLINICAL TRIAL: NCT02817854
Title: Procalcitonin REveals Good Recovery After Acute Diverticulitis: the PREGRAD Study
Brief Title: PCT REveals Good Recovery After Acute Diverticulitis: the PREGRAD Study
Acronym: PREGRAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Valentina Giaccaglia, Valentina Giaccaglia, MD, University of Roma La Sapienza
Other Study IDs: PREGRAD
Record Dates: First submitted 2016-06-27; First posted 2016-06-29 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Acute Diverticulitis
MeSH Terms: interventions — Leukocyte Count; C-Reactive Protein

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with acute diverticulitis: Patients admitted in emergency setting for acute diverticulitis
  Interventions: Procedure: Measure PCT, CRP and WBC at admission; Procedure: Measure PCT, CRP and WBC 1 day after admission; Procedure: Measure PCT, CRP and WBC 2 days after admission

INTERVENTIONS:
Procedure: Measure PCT, CRP and WBC at admission — Measure PCT, CRP and WBC at admission after diagnosis of acute diverticulitis with CT scan has been done
  Other Names: PCT: procalcitonin; WBC: white blood cell count; CRP: C- reactive protein
Procedure: Measure PCT, CRP and WBC 1 day after admission — Measure PCT, CRP and WBC at one day after admission for acute diverticulitis
  Other Names: PCT: procalcitonin; CRP: C- reactive protein; WBC: white blood cell count
Procedure: Measure PCT, CRP and WBC 2 days after admission — Measure PCT, CRP and WBC at 2 days after admission for acute diverticulitis
  Other Names: PCT: procalcitonin; CRP: C- reactive protein; WBC: white blood cell count

SUMMARY:
Diverticular disease is a common disease in developed countries, affecting 2.5 million individuals in the United States (US). Prevalence of diverticula increases with age and goes up to 50 to 66% in patients older than age 80 years. Approximately 10 to 25% of patients with diverticulosis will develop diverticulitis. Acute diverticulitis (AD) accounts for 312,000 admissions and 1.5 million days of inpatient care in the US, where its annual treatment costs exceed 2.6 billion dollars. With the ageing of global population these numbers are expected to rise.

Procalcitonin (PCT) is a biomarker widely used to monitor bacterial infections and guide antibiotic therapy in Intensive Care Units and has been shown to be useful in different surgical fields such as acute appendicitis. Recently, has been demonstrated that PCT and CPR have good predictive value of anastomotic leak (AL) after colorectal surgery.

A multicentric study has been designed to test if PCT, CRP and WBC values might be able to predict the outcomes of patients admitted in emergency setting for acute diverticulitis. In particular if they might distinguish between patients needing only conservative (nothing per os, iv fluids and antibiotics) or interventional therapy such as radiological drain or even surgery, in the aim to optimize and individualize each patients therapy and speed patients discharge.

ELIGIBILITY:
Inclusion Criteria:

* all patients admitted for acute diverticulitis in emergency setting
* with CT scan performed and Hinchey > or = 2

Exclusion Criteria:

* age < 18 years
* pregnant women
* patients with acute diverticulitis without CT scan
* patients with acute diverticulitis with Hinchey I

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted for acute diverticulitis in emergency setting, with CT scan performed
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Need to surgery at 30 days after admission | 1 year

SECONDARY OUTCOMES:
Need of percutaneous drainage | 1 year
Length of hospital stay | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Giaccaglia, MD, Principal Investigator — Sant'Andrea University Hospital, Sapienza Univeristy of Rome
Locations (4):
- Department of Digestive Surgery, University Hospital, Dijon, France
- Italy (3):
  - General and Emergency Surgery, Niguarda Hospital, Milan
  - Department of Surgical and Medical Sciences and Translational Medicine, General Surgery and Emergency Surgery Units, Sant'Andrea Hospital, 'Sapienza' University of Rome, Rome
  - Department of Surgery, General Surgery Unit, Azienda Ospedaliero- Universitaria 'Ospedali Riuniti di Trieste', Trieste

IPD SHARING:
Plan to Share IPD: No